CLINICAL TRIAL: NCT04104659
Title: Multicenter Study of Tau Imaging With the Use of [18F]MK-6240 Tracer in Individuals at Risk for and With Autosomal Dominant Alzheimer's Disease
Brief Title: Study of Tau Imaging With the Use of [18F]MK-6240 Tracer
Acronym: MKADAD
Status: Enrolling by invitation | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology and Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: IRB #201901045
Record Dates: First submitted 2019-04-17; First posted 2019-09-26 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease
Keywords: tau; PET; MK 6240; ADAD
MeSH Terms: conditions — Alzheimer Disease; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MK 6240
  Interventions: Drug: MK 6240

INTERVENTIONS:
Drug: MK 6240 — PET tracer, [18F]MK-6240 (an[18F]tau imaging agent,CerveauTechnologies)that has high affinity for the human phosphorylated tau deposits in AD brain offers new opportunities to investigate tau pathology.(Hostetler, Walji et al. 2016, Lohith, Bennacef et al. 2016, Walji, Hostetler et al. 2016, Lohith, Bennacef et al. 2017, Neelamegam, Yokell et al. 2017).We will evaluate this imaging agent in individuals from families with a known Autosomal Dominant Alzheimer's Disease (ADAD) mutation.
  The planned dosage for [18F]MK-6240 is a single intravenous bolus injection of 185 MBq (5.0 mCi) in a large peripheral vein followed by a 10 mL normal saline (0.9% NaCl) flush.

SUMMARY:
The recent development of a PET tracer,[18F]MK-6240(an[18F]tau imaging agent,CerveauTechnologies)that has high affinity for the human phosphorylated tau deposits in AD brain offers new opportunities to investigate tau pathology. The investigators will evaluate this imaging agent in individuals from families with a known Autosomal Dominant Alzheimer's Disease (ADAD) mutation. This study of tau PET using [18F]MK-6240 is performed in conjunction with DIAN and DIAN Extended Registry (DIAN-EXR).

ELIGIBILITY:
Inclusion Criteria:

1. Participants have met all eligibility criteria for enrollment into the Dominantly Inherited Alzheimer's Network (DIAN) and DIAN Extended Registry (DIAN EXR) study enrollment criteria.
2. Male or female participants, at least 18 years of age.
3. Cognitively normal, or with mild dementia, as assessed clinically.
4. Participant is able and willing to undergo testing (magnetic resonance imaging (MRI)or computed tomography (CT), PET, radioactive tracer injection; forthose unable to undergo MRI, CT will be used to generate regions-of interest).
5. Pre-menopausal women will undergo a urine pregnancy test within 24 hours of drug administration. -

Exclusion Criteria:

1. Has any condition that, in the Investigator's opinion, couldincrease risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants with severechronic back pain might not be able to lie still duringthe scanning procedures).
2. Is deemed likely unable to perform the imaging procedures for any reason.
3. Has hypersensitivity to [18F]MK-6240or any of its excipients.
4. Contraindications to PET, PET-CT or MR(e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate.
5. Severe claustrophobia.
6. Women who are currently pregnant or breast-feeding, and women who do not agree to use reliable contraception, or to refrain from sexual activity for 24 hours following administration of the [18F]MK-6240injection will be excluded from the study.
7. Currently participating in any research studyreceiving an active study medication for AD, an investigational drug, device, imaging, or placebo within the past 30 days before screening, and throughout this clinical trial up to 2-weeks past any study-related procedures.
8. Other than the DIAN study, current or recent (within 12 months prior to screening) participation in research studies involving radioactive agents such that the total research-related radiation dose to the participant in any given year would exceed the limits set forth in the US Code of Federal Regulations (CFR) Title 21 Section 631.1. http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfcfr/CFRSearch.cfm?FR=361.1. It is the responsibility of each site to confirm the date of the most recent PET scan and to work within the guidelines of the local Radioactive Drug Research Committee (RDRC) regarding the imaging interval. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants have met all eligibility criteria for enrollment into the Dominantly Inherited Alzheimer's Network (DIAN) and DIAN Extended Registry (DIAN EXR) study enrollment criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Study the temporal dynamics of tau deposition (using [18F]MK-6240). | 12 years from enrollment
  Aim 3 multivariate linear regression models will be implemented within the general linear mixed model framework and estimated using restricted maximum likelihood estimation. This approach allows for the estimation of the association between [18F]MK-6240 and tauopathy measures across all brain regions to be studied in a single model, by considering the dependency in the plaque measures caused by multiple brain regions being nested within a single patient.
Study the temporal dynamics of tau deposition (using [18F]MK-6240). | 12 years from enrollment
  We will first fit a model in training samples and then use the fitted model to predict the longitudinal changes in tau PET and compare the predicted changes with observed data in independent validation samples. This process will be repeated multiple times, thus correcting for the upward bias and computing "honest" measures of replicability of a specific statistical model. We will repeat the cross-validation process for all scientifically interpretable candidate models that we will consider when comparing to tau PET data. A pseudo-panel from additional cross-sectional datasets can also be used in which observations of different subjects in different time-to-onset lengths are matched across observable covariates.
Study the temporal dynamics of tau deposition (using [18F]MK-6240). | 12 years from enrollment
  A statistical approach will be applied but will consider both Aβ and tau PET. Neuropsychometric measures will be grouped into composites representing working memory, episodic memory, language function, and a global composite. Linear mixed effects models will be implemented including family and DIAN site as random effects. Models will include baseline levels of Aβ PET and tau PET from summary measures, EYO, group (asymptomatic and symptomatic), and all interactions
Study the spatial (both local and distributed) changes of tau deposition (using [18F]MK-6240). | 12 years from enrollment
  Using novel mathematical models, we will correlate the topography of tau PET with both cross-sectional and longitudinal spatial patterns seen with other imaging biomarkers (Aβ PET and MRI [structuraland functional]).
Study the relationship between in vivo tau deposition and neuropathology. | 12 years from enrollment
  We will perform quantitative measures of cortical tauopathy NFT, NP, and neuropil thread (NT) burden in twenty-five brain areas using tau-immunostained sections and automated stereological methods.
Study the relationship between in vivo tau deposition and neuropathology. | 12 years from enrollment
  Neuropathological results will be aligned with in vivo imaging using an ex vivo MRI prior to sectioning.

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be maintained at Washington University. This de-identified data may also be shared with other investigators doing research in similar fields such as Alzheimer disease, other neurological disorders or related brain diseases andabnormalities. These investigators may be at Washington University or at other research institutions. This de-identified data may also be shared with large repositories for broad sharing with the research community. If the participant's research data is placed in one of these repositories, only qualified researchers who have received prior approval from individuals that monitor the use of the datawill be able to look at this information. Information from this research study has been or will be entered into a clinical trial databank that is maintained by the National Institutes of Health/National Library of Medicine.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
URL: http://www.dian-info.org